CLINICAL TRIAL: NCT07147348
Title: A Phase I/II, First-in-human, Open-label, Dose Escalation and Indication Expansion Study of the Safety, Tolerability, Pharmacokinetics, Immunogenicity and Preliminary Efficacy of BNT3212 as Monotherapy or in Combination With BNT327 in Adults With Advanced Solid Tumors
Brief Title: A First-in-human, Dose Escalation and Indication Expansion Study of BNT3212 as Monotherapy or in Combination With BNT327 in Adults With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Biotheus (Hengqin) Co., Ltd. (Unknown); BioNTech (Shanghai) Pharmaceuticals Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BNT3212-01
Record Dates: First submitted 2025-08-08; First posted 2025-08-29 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumor
Keywords: BNT3212 (or PM1300); BNT327; Programmed death-ligand 1 (PD-L1); Vascular endothelial growth factor A (VEGF-A); Bispecific antibody; Antibody-drug conjugate (ADC); Combination with other investigational agents; Immunotherapy; Antibody; Programmed death 1 (PD-1)
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Part A - BNT3212 monotherapy (dose escalation) (Experimental): Escalating dose levels of BNT3212 to define the maximum tolerated dose (MTD) in participants with histologically or cytologically confirmed locally advanced/unresectable, recurrent, or metastatic malignant solid tumors who are refractory to or unable to tolerate standard treatment, or for whom no standard treatment is available.
  Interventions: Biological: BNT3212
- Part B - BNT3212 monotherapy dose level (DL)1 (expansion cohort) (Experimental): Indication-specific cohort populations will be tested.
  Interventions: Biological: BNT3212
- Part B - BNT3212 monotherapy DL2 (expansion cohort) (Experimental): Indication-specific cohort populations will be tested.
  Interventions: Biological: BNT3212
- Part B - BNT3212 monotherapy DL3 (expansion cohort) (Experimental): Indication-specific cohort populations will be tested.
  Interventions: Biological: BNT3212
- Part C - BNT3212 + BNT327 combination therapy (dose escalation) (Experimental): Escalating dose levels of BNT3212 plus a fixed dose of BNT327 to define the MTD in participants with histologically or cytologically confirmed locally advanced/unresectable, recurrent, or metastatic malignant solid tumors who are refractory to or unable to tolerate standard treatment, or for whom no standard treatment is available.
  Interventions: Biological: BNT3212; Biological: BNT327
- Part D - BNT3212 DL1 + BNT327 combination therapy (expansion cohort) (Experimental): Indication-specific cohort populations will be tested.
  Interventions: Biological: BNT3212; Biological: BNT327
- Part D - BNT3212 DL2 + BNT327 combination therapy (expansion cohort) (Experimental): Indication-specific cohort populations will be tested.
  Interventions: Biological: BNT3212; Biological: BNT327
- Part D - BNT3212 DL3 + BNT327 combination therapy (expansion cohort) (Experimental): Indication-specific cohort populations will be tested.
  Interventions: Biological: BNT3212; Biological: BNT327

INTERVENTIONS:
Biological: BNT3212 — Intravenous infusion
Biological: BNT327 — Intravenous infusion
  Arms: Part C - BNT3212 + BNT327 combination therapy (dose escalation); Part D - BNT3212 DL1 + BNT327 combination therapy (expansion cohort); Part D - BNT3212 DL2 + BNT327 combination therapy (expansion cohort); Part D - BNT3212 DL3 + BNT327 combination therapy (expansion cohort)

SUMMARY:
The aim of this first-in-human (FIH) open-label, multi-site study is to evaluate safety, tolerability, pharmacokinetics (PK), immunogenicity and preliminary clinical efficacy of BNT3212, including identification of the recommended dose of BNT3212 for use as monotherapy and with BNT327 as combination therapy, in adults with advanced solid tumors who have exhausted other treatment options.

DETAILED DESCRIPTION:
This study will include four parts (i.e., Parts A, B, C, and D) and follow a stepwise approach, beginning with a typical dose escalation in advanced solid tumors, followed by dose expansion in a range of indications. This design allows to gradually assess safety, preliminary efficacy, potential recommended Phase 2 dose (RP2D), and indications, while ensuring an acceptable benefit-risk balance along the way. Throughout this process, clinical data - including PK, biomarker, immunogenicity, safety, and efficacy, as well as non-clinical data, will be continuously collected and evaluated to support decision-making and ensure participant safety.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants with histologically or cytologically confirmed locally advanced, recurrent, or metastatic solid tumors that have progressed after at least one available standard therapy; or for whom the standard therapy is considered inappropriate or intolerable.
* Have at least one measurable lesion based on RECIST v1.1.
* Eastern Cooperative Oncology Group performance status of 0 (fully active, able to carry out all pre-disease activities without restriction) or 1 (unable to perform physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature).
* Predicted life expectancy of ≥3 months.
* Left ventricular ejection fraction ≥50% by either echocardiography or multigated acquisition scan within 28 days prior to first dose of study treatment.
* Adequate liver, renal, hematological, and coagulation function.
* Recovery to Grade 0-1 (or baseline) from adverse reactions related to prior anti cancer therapy except for:

  * Asymptomatic laboratory abnormalities such as elevated alkaline phosphatase, hyperuricemia, elevated serum amylase/lipase, and elevated blood glucose.
  * Toxicity that the investigator determined to have no safety risk, such as alopecia, Grade 2 peripheral neurotoxicity, hypothyroidism stabilized by hormone replacement therapy, etc.
* The investigator considers discontinuation of protocol-defined anti-cancer therapies and restricted medications with protocol-defined washout periods as medically acceptable.
* For Parts B and D only: Participants must be diagnosed with specific indications.

Key Exclusion Criteria:

* Active infection (e.g., bacterial or fungal infections) requiring systemic treatment (e.g., severe pneumonia, bacteremia, sepsis), except oral antibiotics.
* Participants with primary central nervous system (CNS) malignancies.
* Active CNS metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms.
* Unstable pleural effusion or ascites requiring thoracentesis or paracentesis within 14 days prior to initiation of study treatment.
* Have active, or a history of, pneumonitis requiring treatment with steroids, or has active, or a history of, interstitial lung disease.
* Clinically significant pulmonary complications.
* History of severe cardiovascular disease.
* Have a history of significant hematologic toxicity to prior lines of therapy, as assessed by investigator, e.g., Grade 4 febrile neutropenia or recurrent/persistent Grade 3 to 4 neutropenia.
* Have active or chronic corneal disorders or with any clinically significant corneal disease that prevents adequate monitoring of drug-induced keratopathy.
* Have uncontrolled hypertension while on antihypertensive medicine or poorly controlled diabetes.
* Concurrent malignancy within 5 years prior to study enrollment. Exceptions: basal cell carcinoma, squamous cell carcinoma of the skin, carcinoma in situ after radical resection.
* Unstable thrombotic event (e.g., deep vein thrombosis, arterial thrombosis, pulmonary embolism).
* Have adverse reactions from prior anti-tumor therapy that have not returned to Grade 1 (graded by NCI CTCAE v5.0 criteria) or below (unless the investigator determines that certain AEs pose no safety risk to participants, such as hair loss, Grade 2 peripheral neuropathy or stable hypothyroidism under hormone replacement therapy) are not eligible for the study.
* For Parts C and D only: Prior treatment with PD-1/L1 and VEGF-A antibody combinations (including bispecific antibodies to PD-1/L1 and VEGF-A).
* For Parts C and D only: Have active, or history of, autoimmune disease with risk of exacerbation following PD-L1 inhibition OR an immune deficiency (e.g., allogeneic hematopoietic stem cell transplantation or organ transplantation). Participants with protocol-specified conditions may be eligible.
* For Parts C and D only: Have serious non-healing wounds, ulcer, or bone fracture.
* For Parts C and D only: Have evidence of major coagulation disorders or other significant risks of hemorrhage.
* For Parts C and D only: Have a history of serious Grade 3 or higher immune-related AEs that led to treatment discontinuation of a prior immunotherapy.
* For Parts C and D only: Have a history of small bowel obstruction requiring hospitalization within the past 3 months prior to the first dose of IMP.
* For Parts C and D only: Have received:

  * anticoagulant therapy for therapeutic purposes (except low molecular weight heparin) within 14 days prior to the first dose of IMP.
  * antiplatelet drugs within 10 days prior to the initiation of study treatment.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Parts A and C - Occurrence of dose limiting toxicities (DLTs) within a participant during the DLT observation period | Until 28 days after first dose of investigational medicinal product (IMP).
  Per cohort.
All parts - Percentage of participants with treatment-emergent adverse events (TEAEs) including Grade ≥3, serious, and fatal TEAEs by relationship | From the time of the first dose of IMP until 90 days after the last dose of IMP, approximately up to 31 months.
  Per cohort. Adverse events (AEs) graded according to the National Cancer Institute Common Terminology Criteria for AEs version 5.0 (NCI CTCAE v5.0).
Parts A and C - Percentage of participants with dose interruptions or discontinuations of study treatment due to TEAEs | From the time of the first until last dose of IMP, approximately up to 31 months.
  Per cohort.
Parts B and D - Percentage of participants with dose interruptions, reductions or discontinuations of study treatment due to TEAEs | From the time of the first until last dose of IMP, approximately up to 31 months.
  Per cohort.

SECONDARY OUTCOMES:
All parts - PK assessment: Maximum concentration (Cmax) derived from serum/plasma concentrations | From predose to 28 days after first dose of IMP.
  Per cohort. For BNT3212 (conjugated antibody, total antibody, and unconjugated iCPT) and for BNT327 if in the combination cohorts, as data permits.
All parts - PK assessment: Area under the concentration-time curve (AUC0-t) derived from serum/plasma concentrations | From predose to 28 days after first dose of IMP.
  Per cohort. For BNT3212 (conjugated antibody, total antibody, and unconjugated iCPT) and for BNT327 if in the combination cohorts, as data permits.
All parts - PK assessment: Minimum concentration (Ctrough) derived from serum/plasma concentrations | From predose until 90 days after the last dose of IMP.
  Per cohort. For BNT3212 (conjugated antibody, total antibody, and unconjugated iCPT) and for BNT327 if in the combination cohorts, as data permits.
All parts - Anti-drug antibody (ADA) prevalence | For up to 90 days from the last dose of IMP.
  Per cohort and by dose level, derived from serum samples. Prevalence defined as the proportion of participants who are ADA positive (either baseline or post baseline), if data permits.
All parts - ADA incidence | For up to 90 days from the last dose of IMP.
  Per cohort and by dose level, derived from serum samples. Incidence defined as the proportion of participants having treatment-emergent ADA, if data permits.
All parts - Objective response rate (ORR) | From first dose of IMP until end of study, approximately up to 31 months.
  Per cohort. ORR defined as the proportion of participants in whom a confirmed complete response (CR) or partial response (PR) (per Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST v1.1] based on the investigator's assessment) is observed as best overall response.
All parts - Disease control rate (DCR) | From first dose of IMP until end of study, approximately up to 31 months.
  Per cohort. DCR defined as the proportion of participants with confirmed CR, PR, or stable disease (SD) (per RECIST v1.1 based on the investigator's assessment) as best overall response.
All parts - Duration of response (DOR) | From first dose of IMP until end of study, approximately up to 31 months.
  Per cohort. DOR defined as the time from first confirmed objective response (CR or PR per RECIST v1.1 based on the investigator's assessment) to first occurrence of objective tumor progression (progressive disease [PD] per RECIST v1.1 based on the investigator's assessment) or death from any cause, whichever occurs first.
All parts - Progression free survival (PFS) | From first dose of IMP until end of study, approximately up to 31 months.
  Per cohort. PFS based on the investigator's assessment defined as the time from first dose of trial treatment to the first objective tumor progression (PD per RECIST v1.1) or death from any cause, whichever occurs first.
All parts - Time to response (TTR) | From first dose of IMP until end of study, approximately up to 31 months.
  Per cohort. TTR, defined as the time from first dose of trial treatment to first confirmed objective response (CR or PR per RECIST v1.1 based on the investigator's assessment) in participants with a confirmed objective response.
All parts - Overall survival (OS) | From first dose of IMP until end of study, approximately up to 31 months.
  Per cohort. OS defined as the time from first dose of trial treatment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (2):
- Scientia Clinical Research Limited, Randwick, Australia
- Shanghai East Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No